CLINICAL TRIAL: NCT02944851
Title: Comparison of Noninvasive Two Methods to Monitoring Blood Loss; Inferior Vena Cava (IVC) Ultrasound - Non-invasive Hemoglobin Measurement (SpHb)
Brief Title: Comparison of the Accuracy of Non-invasive Hemoglobin Measurement (SpHb) and Vena Cava Inferior Ultrasound
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Emergency medicine specialist, Emergency Department, Haseki Training and Research Hospital
Other Study IDs: 336
Record Dates: First submitted 2016-09-26; First posted 2016-10-26 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Blood Donors, Traumatic Blood Loss
Keywords: Blood donors; blood donation; traumatic blood loss; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective observational: The changes of IVC diameter, SpHb and vital signs of blood donors were observed after blood donation

SUMMARY:
The aim of this work is determine the more successful noninvasive method by comparison of two noninvasive methods ( IVC ultrasound - noninvasive hemoglobin measurement (SpHb)) that used in the detection of patients with blood loss.

The works were completed in 6 months. The study was conducted at the blood donation center and in Emergency department. Vital parameters were measured and recorded before making the voluntary blood donation. Following Masimo brand portable device fingers SpHb value was measured.Then IVC diameter of patients in the supine position were measured using ultrasonography. Then he left to donors return in routine blood donation programme. A unit (500ml) of blood were drawn from each donor. After the blood donation process measured and recorded the vital signs again. SpHb was measured noninvasively from finger again. Following these measurements were recorded again by measuring the diameter of IVC.

ELIGIBILITY:
Inclusion Criteria:

* Who have volunteered to donate blood
* Older than 18 years
* Both sexes

Exclusion Criteria:

* Known tricuspid valve regurgitation and right heart failure
* Oral intake or the fluid loss (diarrhea and vomiting-urination) between the two measurements during the blood donation
* Inappropriate echogenicity for vena cava inferior diameter measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voluntary donors for blood donation.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of stage 1 hemorrhagic shock | 30 minute (15 minute blood donation, 15 minute rest time ).
  Changes in IVC diameter were observed with 500 ml blood loss. Measurement were made pre and post blood donation.
Diagnosis of stage 1 hemorrhagic shock | 30 minute (15 minute blood donation, 15 minute rest time ).
  Changes in SpHb were observed with 500 ml blood loss. Measurement were made pre and post blood donation.

SECONDARY OUTCOMES:
Diagnosis of stage 1 hemorrhagic shock | 30 minute (15 minute blood donation, 15 minute rest time ).
  Changes in Pulse rate were observed with 500 ml blood loss. Measurement were made pre and post blood donation.
Diagnosis of stage 1 hemorrhagic shock | 30 minute (15 minute blood donation, 15 minute rest time ).
  Changes in Arterial blood pressure were observed with 500 ml blood loss. Measurement were made pre and post blood donation.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Yamanoğlu, MD, Study Director — The health ministry, Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Reseurch Hospital, Istanbul, Turkey (Türkiye)